CLINICAL TRIAL: NCT03296059
Title: Transfusion of Red Blood Cells for Acute Respiratory Distress Syndrome(ARDS) in Neonates: A Randomized Controlled Trial
Brief Title: Transfusion of Red Blood Cells for Acute Respiratory Distress Syndrome(ARDS) in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ma Juan, director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201732
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Red Blood Cells(RBC); Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RBC transfusion with conventional treatment (Experimental): Besides conventional treatment,neonates diagnosed with ARDS is treated with RBC transfusion.
  Interventions: Other: conventional treatment with RBC transfusion
- conventional treatment (Active Comparator): neonates diagnosed with ARDS is treated with conventional treatment.
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: conventional treatment with RBC transfusion — Besides conventional treatment, neonates is given RBC transfusion.
  Arms: RBC transfusion with conventional treatment
Other: conventional treatment — neonates is treated with conventional treatment.
  Arms: conventional treatment

SUMMARY:
Acute respiratory distress syndrome (ARDS) in neonates has been defined in 2017.

The death rate is over 50%.There are no special treatments for acute respiratory distress syndrome.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is one of the serious complications in critically ill neonates. It can result in severe hypoxemia refractory to mechanical ventilation. There are few options for mechanical ventilation for such situations such as high frequency oscillation ventilation and extracorporeal membrane oxygenation. The aim of the present study is to determine whether transfusion of red blood cells can decrease the mortality in neonate with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with neonatal ARDS.
* informed parental consent has been obtained

Exclusion Criteria:

* major congenital malformations or complex congenital heart disease
* transferred out of the neonatal intensive care unit without treatment

Ages: 30 Minutes to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
death rate | within 100 days
  neonate died due to respiratory failure

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066